CLINICAL TRIAL: NCT00877058
Title: Elderly Persons at the Risk Zone - a Randomized Controlled Trial of a Community Based Preventive Multiprofessional Program for Old Persons at Risk of Frailty
Brief Title: SUPPORT FOR FRAIL ELDERLY PERSONS - From Prevention to Palliation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Responsible Party: Principal Investigator, Synneve Dahlin Ivanoff, Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: G213 194/08
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Frail Elderly Persons
Keywords: Frailty; health promotion; prevention; self management; intervention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.Preventive home visit (Experimental): Preventive home visits: This intervention included a single home visit made by either a nurse, a physiotherapist, a qualified social worker or an occupational therapist. Participants received verbal and written information/advice about what the districts could provide. The preventive home visit was guided by a protocol, which included an opportunity for individuals to further elaborate on certain elements. The visit lasted between one and a half to two hours.
  Interventions: Behavioral: preventive home visit
- 2. Senior meetings (Experimental): The senior meetings comprised four weekly meetings with about six participants in each group. The main purpose was to focus on two different topics: 1) information about the ageing process and its consequences and 2) provision of tools and strategies for solving problems that can arise in the home environment. A follow-up home visit took place two to three weeks after the group sessions were completed. The group meetings were led either by an occupational therapist, a registered nurse, a physiotherapist or a qualified social worker, all of whom spoke about their particular dimension of aging.
  Interventions: Behavioral: senior meetings
- 3. Control group (No Intervention): The control group had access to the ordinary range of services if requested from the urban districts for the aged. The aim of the municipal provision of care for the older persons is to ensure the ability to live as independently as possible. This includes remaining in their homes. When an older person in Sweden has difficulties managing independently, she or he can apply for assistance from the district. The extent of such support is subject to an assessment of needs and includes meals on wheels, help with cleaning and shopping, assistance with personal care, safety alarms and transportation service. The older person are also offered healthcare, provided either by municipal home help or home medical care services.

INTERVENTIONS:
Behavioral: preventive home visit
  Arms: 1.Preventive home visit
Behavioral: senior meetings
  Arms: 2. Senior meetings

SUMMARY:
The present study "Elderly person in the risk zone" form part of the research programme "Support for frail elderly persons - from prevention to palliation" (www. Vardalinstitutet.net) which comprises research into three interventions. A fundamental principle in the research programme is that it comprises interventions addressing frail elderly person in different phases of the disablement process, from elderly persons who are beginning to develop frailty to very frail elderly persons receiving palliative care in the final period of their lives. The interventions also address the different requirements that arise with regard to professional contributions during the various phases of the ageing and disease process, ranging from health promotion to a need for an increasing degree of medical care, nursing, special care and rehabilitation, and finally, efforts that promote symptom relief, quality of life, security and satisfaction with care during the final period of life. The intervention "Elderly persons in the risk zone" addresses elderly persons that are on the point of developing frailty ("pre-frail") and are beginning to feel that they are being hindered from taking part in everyday activities. The hypothesis is that if an intervention is made when the persons are not so frail, it is possible to prevent/delay deterioration.

1. Can a health-promoting and preventive intervention for "prefrail" elderly persons:

   * prevent frailty, activity limitations and morbidity,
   * be a supportive factor in the social and physical environment,
   * affect life satisfaction
   * have an impact on the consumption of care
   * be cost-effective?
2. How do the frail elderly persons experience the intervention and its importance to health?

ELIGIBILITY:
Inclusion Criteria:

* 80 years of age or older living in the community.
* The participants should live in their ordinary housing
* Independent on formal support
* Independent on informal support
* Cognitive intact defined as a Mini Mental Test score > 25

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 459 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Synneve Dahlin Ivanoff, Professor, Principal Investigator — Göteborg University
Locations (1):
- Gothenburg University, Gothenburg, Sweden

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Dahlin-Ivanoff S, Eklund K, Wilhelmson K, Behm L, Haggblom-Kronlof G, Ziden L, Landahl S, Gustafsson S. For whom is a health-promoting intervention effective? Predictive factors for performing activities of daily living independently. BMC Geriatr. 2016 Oct 6;16(1):171. doi: 10.1186/s12877-016-0345-8. PMID 27716095
- [Derived] Dahlin-Ivanoff S, Gosman-Hedstrom G, Edberg AK, Wilhelmson K, Eklund K, Duner A, Ziden L, Welmer AK, Landahl S. Elderly persons in the risk zone. Design of a multidimensional, health-promoting, randomised three-armed controlled trial for "prefrail" people of 80+ years living at home. BMC Geriatr. 2010 May 26;10:27. doi: 10.1186/1471-2318-10-27. PMID 20504358

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Preventive Home Visits: This intervention included a single home visit made by either a nurse, a physiotherapist, a qualified social worker or an occupational therapist. Participants received verbal and written information/advice about what the districts could provide. The preventive home visit was guided by a protocol, which included an opportunity for individuals to further elaborate on certain elements. The visit lasted between one and a half to two hours.
- 2 Senior Meetings: The intervention senior meetings comprised four weekly meetings with about six participants in each group. The main purpose was to focus on two different topics: 1) information about the ageing process and its consequences and 2) provision of tools and strategies for solving problems that can arise in the home environment. A follow-up home visit took place two to three weeks after the group sessions were completed. The group meetings were led either by an occupational therapist, a registered nurse, a physiotherapist or a qualified social worker, all of whom spoke about their particular dimension of aging. They jointly planned and carried out the intervention and were responsible for their specific part of the meetings. T The participants' experiences formed the basis of the meetings. A booklet was especially produced for the meetings, which includes texts that cover different areas of health, discussed at each of the meetings. http://www.vardalinstitutet.net/livslots.pdf.
- 3 Control Group: The control group had access to the ordinary range of services if requested from the urban districts for the aged. The aim of the municipal provision of care for the older persons is to ensure the ability to live as independently as possible. This includes remaining in their homes. When an older person in Sweden has difficulties managing independently, she or he can apply for assistance from the district. The extent of such support is subject to an assessment of needs and includes meals on wheels, help with cleaning and shopping, assistance with personal care, safety alarms and transportation service. The older person are also offered healthcare, provided either by municipal home help or home medical care services.
Period: Overall Study
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group
Started | 174 | 171 | 114
Completed | 137 | 131 | 75
Not Completed | 37 | 40 | 39

BASELINE CHARACTERISTICS:
Groups:
- 2 Senior Meetings: The intervention senior meetings comprised four weekly meetings with about six participants in each group. The main purpose was to focus on two different topics: 1) information about the ageing process and its consequences and 2) provision of tools and strategies for solving problems that can arise in the home environment. A follow-up home visit took place two to three weeks after the group sessions were completed. The group meetings were led either by an occupational therapist, a registered nurse, a physiotherapist or a qualified social worker, all of whom spoke about their particular dimension of aging. They jointly planned and carried out the intervention and were responsible for their specific part of the meetings. T The participants' experiences formed the basis of the meetings. A booklet was especially produced for the meetings, which includes texts that cover different areas of health, discussed at each of the meetings (table 1). http://www.vardalinstitutet.net/livslots.pdf.
- Total: Total of all reporting groups
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group | Total
Number analyzed (Participants) | 174 | 171 | 114 | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 174 | 171 | 114 | 459
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  ≥80 years | 86 [80 to 97] | 85 [80 to 94] | 86 [80 to 97] | 86 [80 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 113 | 70 | 294
  Male | 63 | 58 | 44 | 165
Region of Enrollment [Number; unit: participants]
  Sweden | 174 | 171 | 114 | 459

OUTCOME MEASURES:

1. Primary Outcome: Dependence in Two or More Activities of Daily Living (ADL)
Description: ADL stair case:
  Independence of, or dependence on, another person in ADL was assessed according to a cumulative scale of well-defined personal and instrumental activities, the ADL staircase. Nine out of the ten original activities were used; Cleaning, shopping, transportation, cooking, bathing, dressing, going to the toilet, transfer, and feeding (0-9). Dependence was defined as another person being involved in the activity by giving personal or directive assistance. People living together were assessed as independent if they performed the activity when alone. The number of partipants with dependence in two or more ADL at follow-up have been analyzed
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group
Number analyzed (Participants) | 174 | 171 | 114
participants | 35 | 26 | 44
Statistical Analysis 1: Comparison: 2 Senior Meetings vs 3 Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.15 to 0.48]
Statistical Analysis 2: Comparison: 1 Preventive Home Visits vs 3 Control Group; Test type: Superiority or Other; p = 0.001, Chi-squared; Odds Ratio (OR) = 0.40, 0.05% CI 2-sided [0.24 to 0.68]

2. Primary Outcome: Number of Partipants Measured Frail at 1-year Follow up
Description: Frailty defined as a sum of weakness, fatigue, weight loss, low physical activity, poor balance, slow gait speed, visual impairment and impaired cognition
Time Frame: 1 year
Population: ITT was used. The basic assumption was that older adults (80+) deteriorate over time in the natural course of the aging process. The imputation method chosen was to replace missing values with a value based on the Median Change of Deterioration (MCD) a conservative form of worst case between baseline and follow-up.
Measure: Number; unit: participants
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group
Number analyzed (Participants) | 174 | 171 | 114
participants | 80 | 85 | 43
Statistical Analysis 1: Comparison: 2 Senior Meetings vs 3 Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.96 to 2.52]
Statistical Analysis 2: Comparison: 1 Preventive Home Visits vs 3 Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.79 to 2.08]

3. Primary Outcome: Self Rated Health
Description: Self rated health was measured by the question "In general would yoy say your health is: excellent, very good, good, fair or poor? Number of participants detoriated in self-rated health has been analysed
Time Frame: 1 year
Population: ITT
Measure: Number; unit: participants
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group
Number analyzed (Participants) | 174 | 171 | 114
participants | 31 | 29 | 31
Statistical Analysis 1: Comparison: 2 Senior Meetings vs 3 Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.31 to 0.97]
Statistical Analysis 2: Comparison: 1 Preventive Home Visits vs 3 Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.33 to 1.02]

ADVERSE EVENTS:
Arm/Group | 1 Preventive Home Visits | 2 Senior Meetings | 3 Control Group
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/171 | 0/114
Other Adverse Events (participants affected / at risk) | 0/174 | 0/171 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No